CLINICAL TRIAL: NCT03313661
Title: Co-administration of Cabergoline and Gliclazide Improve Glycemic Parameters and Lipid Profile in T2DM Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diabetes Mellitus
Record Dates: First submitted 2017-10-14; First posted 2017-10-18 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Cabergoline; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cabergoline (Experimental): cabergoline 0.5 mg twice weekly within 2 hrs of awakening plus gliclazide
  Interventions: Drug: Cabergoline
- Gliclazide (Active Comparator): gliclazide (60-120 mg) once daily
  Interventions: Drug: Gliclazide
- Placebo (No Intervention): Placebo

INTERVENTIONS:
Drug: Cabergoline — cabergoline 0.5 mg twice weekly within 2 hrs of awakening plus gliclazide
  Arms: Cabergoline
Drug: Gliclazide — gliclazide (60-120 mg)
  Arms: Gliclazide

SUMMARY:
Evaluation of the glycemic efficacy of cabergoline on diabetic patients

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (DM) is a progressive metabolic disorder that is associated with basal hyperinsulinemia, insulin resistance and impaired insulin release. Glycemic control is a fundamental part of the management of type 2 DM and difficult to achieve. Different antidiabetic agents can handle diabetic metabolic abnormalities. The development of antidiabetic agentswith novel mechanisms of action is highly desirable. Cabergoline, a long acting D2 agonist, is expected to play a role in the glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients.

Exclusion Criteria:

* Other drugs administration

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-14 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The level of fasting and post prandial BG level | 4 months
  Fasting and post prandial BG level will be measured after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jouliana Atef Morcos, Msc, Study Chair — Faculty of Pharmacy, Tanta University, Egypt; Abla Mohamed Ebeid, Ph D, Study Chair — Faculty of Pharmacy, AL-Delta University, Gamasa, Egypt; Samy Abdel kader khodeir, Ph D, Study Chair — Tanta University; Gamal Abdel khalek Elazab, Ph D, Study Chair — Faculty of Pharmacy, Tanta University, Egypt
Locations (1):
- Sherief Abd-Elsalam, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided